CLINICAL TRIAL: NCT07342101
Title: A Multicenter, Prospective, Randomized, Double-Blind, Open-Label Clinical Trial Evaluating the Effects of Lacticaseibacillus Rhamnosus GG on Acute Infectious Diarrhea in Children in Türkiye
Brief Title: Evaluating the LGG of on Acute Infectious Diarrhea in Children
Acronym: PROBAGE 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ener Cagri DINLEYICI, Professor in Pediatrics, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROBAGE-V0-2025-12
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Acute Infectious Diarrhoea in Children
Keywords: probiotic; diarrhea; LGG
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): LGG with standart of care
  Interventions: Other: LGG; Other: Standart of care
- Control (Active Comparator): Standart of care
  Interventions: Other: Standart of care

INTERVENTIONS:
Other: LGG — Lacticaseibacillus rhamnosus GG 5 billion CFU, twice daily for 6 days
  Arms: Probiotic
Other: Standart of care — ORS (depends on body weight) and/or intravenous fluids

SUMMARY:
Acute diarrhea due to infectious causes is a major source of morbidity in the pediatric population.

Although it is generally self-limiting, acute diarrhea may lead to severe dehydration, hospitalization, and, rarely, death, particularly in young children. Numerous studies have investigated the role of probiotics and other microbiota-targeted therapies in improving the clinical course of infectious acute diarrhea.

The first multicenter PROBAGE study conducted in Türkiye 15 years ago provided valuable evidence regarding the efficacy of probiotics in this context. Over the past 15 years, changes in epidemiology-especially in the post-pandemic period-have created a need for new studies evaluating the effectiveness of probiotics in acute diarrhea.

The PROBAGE 2.0.1 study is designed to evaluate the efficacy of Lactobacillus rhamnosus GG in the treatment of acute infectious diarrhea in children in Türkiye. This is a multicenter, prospective, randomized, open-label, controlled clinical trial, to be conducted across seven tertiary care medical centers nationwide. A total of 480 children with acute infectious diarrhea will be enrolled.

At the initial presentation, stool samples will be collected to identify rotavirus, norovirus, and adenovirus as causative pathogens. The treatment group (n = 240) will receive standard of care plus Lactobacillus rhamnosus GG (one sachet twice daily for 5 or 10 days), whereas the control group (n = 240) will receive standard of care alone.

Daily monitoring of stool frequency and consistency will be documented for 10 days, by families for outpatients and by physicians and nurses for hospitalized patients. Provided that sufficient data are obtained, data analysis and publication phases will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month to 10 years presenting with acute infectious diarrhea (for S. boulardii group)
* Children aged 2 to 10 years presenting with acute infectious diarrhea (other probiotics or synbiotics groups)
* Onset of diarrhea symptoms within the last 48 hours.
* Parental/legal guardian consent obtained.

Exclusion Criteria:

* Use of any probiotics or biotic formulations within the past 8 weeks.
* Use of antibiotics in the last 8 weeks.
* Presence of chronic diseases (e.g., diabetes, congenital heart disease, immunodeficiencies).
* Previous gastrointestinal surgical procedures.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
duration of diarrhea | 10 days
  Mean duration of diarrhea (in days), defined as the time from onset until the return to normal stool consistency and frequency.

SECONDARY OUTCOMES:
Proportion of diarrhea cases lasting >5 days | 5 days

IPD SHARING:
Plan to Share IPD: No